CLINICAL TRIAL: NCT03850041
Title: The Variability and Impact of Segmental Neck and Leg Fluid Volume Shifts on Upper Airway Collapse and Obstructive Sleep Apnea (OSA) Severity in Surgical Patients With OSA
Brief Title: The Impact of Fluid Volume Shifts on Upper Airway Collapse and Obstructive Sleep Apnea in Surgical Patients
Status: Terminated | Type: Observational
Why Stopped: lapse of renewal
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Lung Association (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-5747
Record Dates: First submitted 2019-01-30; First posted 2019-02-21 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to examine the contribution of intravenous (IV) fluid administration and rostral fluid shift from the legs to the neck thereby leading to worsening of sleep apnea following surgery. In this prospective, observational cohort study, 50 consecutive preoperative adult obstructive sleep apnea (OSA) patients, requiring at least one night hospital stay post surgery, will be recruited. Recent research from general population suggests that intravenous (IV) fluid administration worsens the severity of OSA by shifting of fluid from the legs to the neck thus increasing neck size and causing airway collapse. The results of this study will be used to design future clinical trials evaluating methods to decrease postoperative OSA worsening, as well as decreasing OSA-related postoperative complications.

DETAILED DESCRIPTION:
The study investigators hypothesize that in obstructive sleep apnea (OSA) patients undergoing elective non-cardiac surgery, preferential increase in neck fluid volume following intravenous administration during general anesthesia results in worsening apnea-hypopnea (AHI) and postoperative respiratory complications.This is a two-center study where the study population will be drawn from patients visiting preoperative clinic at University Health Network Hospitals, Toronto Western Hospital, and Toronto General Hospital.

Objectives of the study

* Measure the change in the leg, neck and total fluid volume from preoperative baseline, postoperative care unit (PACU), first postoperative night (Night 1) and the morning after surgery (Day 2)
* Assess the impact of the change in neck fluid volume on respiratory mechanics and postoperative apnea-hypopnea index (AHI) the first postoperative night (Night 1) In this study, the investigators will perform serial measurements of segmental and total body water shifts occurring after surgery, at various time-points on the night and the morning after surgery. The investigators will monitor indices such as the Apnea Hypopnea index (AHI) and oxygen desaturation index (ODI) to examine changes in the severity of OSA. Internal validity of this study will be made more robust by use of well-validated methods such as Bioelectrical Impedance Analysis (BIA) for fluid measurements, portable Apnea Link for OSA severity and tremflow airway oscillometry for the airway resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 yrs)
2. Previously diagnosed OSA (AHI > 10), untreated or non-compliant to treatment, or patients screened as suspected OSA (STOP Bang >3, and confirmed to have OSA with AHI > 10 on a portable sleep study)
3. ASA physical status I - IV
4. Patients undergoing elective non-cardiac surgery under general anesthesia;
5. Patients requiring overnight admission.

Exclusion Criteria:

1. Patients compliant on OSA treatment such as continuous positive airway pressure therapy or an oral appliance
2. Vascular surgery on the lower limbs, or metal implants in lower limbs
3. Pregnant or lactating patients
4. Cardiac, intra-cranial, or neck procedures.
5. Inability to communicate: with health care providers or the research personnel, inability to perform breathing maneuvers such as spirometry, or inability to follow instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients attending the preoperative assessment clinic in Toronto Western Hospital (UHN) who will be undergoing elective non-cardiac surgery, requiring general anesthesia, lasting for 1-2 hours or more and requiring same day admission for a minimum of 2 days postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Neck, leg and total body water volumes preoperatively and on postoperative night 1 and the morning after surgery | 24 hours
  Measurement of the leg fluid, neck fluid and total body water using the bioelectrical impedance analysis.
Apnea-hypopnea index on the night of surgery | 24 hours
  Measurement of the AHI (Apnea-hypopnea index) events/hour ,to determine severity of Obstructed Sleep Apnoea on the night of the surgery, using the following scale for ApneaLink device data:
  1. No OSA( AHI: 0-5 events/hour),
  2. Mild OSA(AHI: 6 to 15 events/hour),
  3. Moderate OSA (AHI : 16-30 events/hour) and
  4. Severe OSA (AHI: >30 events/hour),

SECONDARY OUTCOMES:
Neck Circumference on Postoperative Night 1 | 24 hours
  Neck circumference (in cm) will be assessed with a measuring tape and reported for correlation with other data

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Result] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Result] Mutter TC, Chateau D, Moffatt M, Ramsey C, Roos LL, Kryger M. A matched cohort study of postoperative outcomes in obstructive sleep apnea: could preoperative diagnosis and treatment prevent complications? Anesthesiology. 2014 Oct;121(4):707-18. doi: 10.1097/ALN.0000000000000407. PMID 25247853
- [Result] Ng SS, Chan TO, To KW, Ngai J, Tung A, Ko FW, Hui DS. Validation of a portable recording device (ApneaLink) for identifying patients with suspected obstructive sleep apnoea syndrome. Intern Med J. 2009 Nov;39(11):757-62. doi: 10.1111/j.1445-5994.2008.01827.x. Epub 2008 Nov 3. PMID 19220528
- [Derived] Lukachan GA, Chung F, Yadollahi A, Auckley D, Eissa M, Rahman N, McCluskey S, Singh M. Perioperative trends in neck and leg fluid volume in surgical patients: a prospective observational proof-of-concept study. Can J Anaesth. 2023 Feb;70(2):191-201. doi: 10.1007/s12630-022-02362-6. Epub 2022 Nov 30. PMID 36450944
- See also: Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. — https://www.ncbi.nlm.nih.gov/pubmed/11254524?dopt=Abstract
- See also: Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. — https://www.ncbi.nlm.nih.gov/pubmed/18431116?dopt=Abstract
- See also: Anesthesiology. 2014 Oct;121(4):707-18. doi: 10.1097/ALN.0000000000000407. A matched cohort study of postoperative outcomes in obstructive sleep apnea: could preoperative diagnosis and treatment prevent complications? — https://www.ncbi.nlm.nih.gov/pubmed/25247853?dopt=Abstract
- See also: Intern Med J. 2009 Nov;39(11):757-62. doi: 10.1111/j.1445-5994.2008.01827.x. Epub 2008 Nov 3. Validation of a portable recording device (ApneaLink) for identifying patients with suspected obstructive sleep apnoea syndrome. — https://www.ncbi.nlm.nih.gov/pubmed/19220528?dopt=Abstract